CLINICAL TRIAL: NCT03630744
Title: Fluid Day: Observational Study About Fluid Therapy Administered in Adult Patients Undergoing Surgery in Our Country
Brief Title: Fluid Day Spanish Observational Study
Acronym: Fluid Day
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sociedad Española de Anestesiología, Reanimación y Terapéutica del Dolor (Other)
Collaborators: Hospital Vall d'Hebron (Other); Hospital Universitario Infanta Leonor (Other); Hospital Verge dels Lliris (Unknown); Hospital Clinic of Barcelona (Other); Hospital Universitario Doctor Peset (Other); Hospital Miguel Servet (Other); Hospital Universitario La Fe (Other)
Responsible Party: Principal Investigator, Maria José Clara Colomina Soler, Principal Investigator, Hospital Universitari de Bellvitge
Other Study IDs: HTF-FLU-2018-01; SED-HEA-2018-01 (Registry Identifier: Spanish agency of medicine and health products)
Record Dates: First submitted 2018-06-30; First posted 2018-08-15 (Actual); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Fluid Therapy
Keywords: fluid theraphy; surgical procedures; adult patients; glycocalyx; practice guideline
MeSH Terms: interventions — Fluid Therapy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult patients undergoing surgery: Patients over 18 years surgically treated with fluid therapy during the 24 hours of the day study
  Interventions: Other: Fluid therapy

INTERVENTIONS:
Other: Fluid therapy — * Analyze the type of fluid administered:
    * crystalloids:
      * Saline serum 0.9% ....... ml
      * Ringer Lactate ........ ml
      * Isofundin ® ........ ml
      * Plasmalyte® ... ... ml
      * Glucose Serum 5% ....... ml
      * Glucose serum 10% ........ ml
    * Glucosaline serum ........ ml
    * colloids:
      * Hydroxyethyl starch 130 / 0.4 ... ... ml
      * Hydroxyethyl alimdon 130 / 0.42 ... .... ml
      * Gelatins ... ....... ml
      * Albumin 5% .......... ml
    * Albumin 20% .......... ml.
  * Analyze the total amount of crystalloids and liquid colloids administered in 24 hours in milliliters.
  * Analyze the form of administration:
    * Standard
    * Standard with dosimeters
    * on pump

SUMMARY:
Perioperative fluid therapy has undergone a huge change in clinical practice in recent years. The patterns of replacement and / or restoration of volemia described in the classic anaesthesiology books were supported by weak scientific evidence, and a paradigm shift in perioperative fluid therapy based on aspects such as increased mortality associated with an excessively positive balance of fluids in the perioperative period, evidences related to the non-existence of the third non-anatomical space and the need to preserve the capillary endothelium and its glycocalyx.

On the other hand, advances in technology, through the availability of less invasive monitoring systems, capable of determining dynamic parameters related to blood volume that allow predicting the response to volume management, have provided much more adequate monitoring and simple to guide such intravenous volume restoration.

Following all these changes different guidelines and recommendations have been published in recent years with the intention of clarifying the current evidence and facilitate the correct use of fluid therapy to clinicians, but despite this the fact is that today the investigators still do not have information on how fluid therapy is administered in daily practice, so the section of Hemostasis, Transfusion Medicine and Fluid Therapy of SEDAR, considered it necessary to evaluate the clinical practice of fluid therapy in the perioperative period through the Fluidday study.

DETAILED DESCRIPTION:
Background: The administration of fluids in the perioperative period is a routine clinical practice that sometimes underestimates the repercussion of its correct administration.

According to the guidelines of the Spanish Society of Anesthesiology, Resuscitation and Therapy of Pain (SEDAR), the objective of perioperative fluid therapy is to maintain the organism with an optimal state of tissue perfusion and hydration.

This goal is not always easy to carry out. The continuous changes in surgical and anesthetic techniques and the appearance of new fluids and monitoring devices make it difficult for the anesthesiologist to carry out all these changes in his daily clinical practice. For this reason, SEDAR and other international scientific societies have recently published guidelines on the management of fluid therapy in the perioperative period, with the intention of facilitating the decision making of the anesthesiologist in their usual clinical practice based on current evidence. Also adding the recent withdrawal and commercial suspension of a special type of fluid such as Hydroxyethylstarch.

Hypothesis: Fluid therapy in the surgical environment is administered in a protocolized manner and in accordance with the recommendations of the different clinical practice guidelines.

Objectives: To evaluate the management of fluid therapy by anesthesiologists in adult patients during the perioperative period of scheduled and urgent surgery, taking into account the types of fluids administered, the monitoring used and the application of guided therapy protocols by objectives.

Methods: A multicenter prospective observational cross-sectional study - 24-hour Prevalence Cut off is proposed to evaluate the fluid therapy administered by anesthesiologists in surgical patients. The study will be carried out simultaneously in all hospitals that decide to participate throughout the Spanish territory and the follow-up period will be a maximum of 24 hours. Two different intersemanial days will be chosen to include the maximum number of episodes and types of surgeries.

Relevance: The clinical practice guidelines with their recommendations or suggestions offer a safety tool for patients based on current scientific evidence, hence the importance of its correct implementation. Sometimes problems of dissemination of information or limitations in the application of the same can cause that these objectives are not met.

From the Section of Hemostasis, Transfusion Medicine and Fluid Therapy of the SEDAR, it is intended to assess the implementation and follow-up of the recommendations and / or suggestions issued in the different clinical practice guidelines for the correct management of Fluid Therapy in the perioperative setting by performing of this study. This will allow locating the points of improvement in the usual clinical practice on perioperative fluid therapy and will contribute on the one hand to the implementation of the different clinical practice guidelines and, on the other hand, it will serve as a base material for the development of future lines of research.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age surgically treated during the 24 hours of the two-day study of both scheduled and emergency surgery.

Exclusion Criteria:

* Interventions performed outside the surgical area: complementary examination cabinets.
* Interventions that do not require the presence of an anesthesiologist.
* Ophthalmologic surgery
* Surgery performed with local anesthesia.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population The fluid therapy administered by the anesthesiologists (Operating Room, PACU and resuscitation and critical units) will be recorded for all patients who are operated during the 24 hours of the study and who meet the inclusion criteria. The 24 hours of registration will be defined as the interval of 08:00 a.m. of the chosen day until 08:00 a.m. of the next day.
  Participation in this study only involves conducting an interview and collecting data from your clinical record referring to the 24 hours after your intervention, without making any additional intervention.
Sampling Method: Non-Probability Sample
Enrollment: 3500 (Estimated)
Dates: Start 2019-02 (Estimated); Primary Completion 2019-02 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Management of fluid theraphy in the operating room and postoperative care. | Two days
  The purpose of this study is to evaluate how fluids are administered in the Operating Room and postoperative care. We also collect data on the total amount of fluids administered and the type of fluid administered during the anesthesia procedure and surgery.
  Type of Crystalloids and total amount in mL
  * Saline serum 0.9% ....... ml
  * Lactated Ringer ........ ml
  * Isofundin ® ........ ml
  * Plasmalyte® ... ... ml
  * Glusose 5% ....... ml
  * Glucose 10% ........ ml
  * Saline & Glucose 5% ........ ml Type of Colloids and total amount in mL
  * HEA 130 / 0.4 ... ... ml
  * HEA 130 / 0.42 ...... .... ml
  * Gelatins ... ....... ml
  * Albumin 5%.......... ml
  * Albumin 20% ………..ml
  Method of administration:
  * Standard
  * Standard with dosimeters
  * In pump Use of goal-guided Fluid Therapy protocols
  * YES
  * NO
  Use of Hemocomponents type and total does in mL:
  * RBC..........mL
  * Plasma..........................ml
  * Platelets ..........ml

SECONDARY OUTCOMES:
Monitorization | Two days
  Type of monitors used in the operating room and postoperative care.
  * Standard (NIBP, ECG, SpO2)
  * Invasive Blood Pressure
  * PVC
  * Advanced hemodynamics: Specify: □ CAP □ TTP □ DTL □ TEE □ COP □ Other
  * Dynamic Preload Parameters: Specify: □ VVS □ VPS □ VPP □ IVP
  Targeted therapy protocol (Yes / No)
  PANI: Non-invasive blood pressure ECG: Electrocardiogram SpO2: Partial oxygen saturation PVC: Central venous pressure CAP: Pulmonary artery catheter GC: Cardiac output TTP: Pulmonary thermodilution DTL: Transpulmonary Lithium Dilution ETT: Transesophageal echocardiography VVS: Systolic volume variation VPS: Systolic pressure variation VPP: Pulse pressure variation IVP: Index of plethysmographic variation
Demographic | Two days
  Sex
  * Female
  * man Age……..years old Weight …….Kg Height ……..cms BMI ASA
Commorbidities | Two days
  Renal Insufficiency
  * Yes
  * No Heart Failure
  * Yes
  * No Cardiac valve disease
  * Yes
  * no Pulmonary Hypertension
  * Yes
  * No Hepatopathy,
  * Yes
  * NO Arterial Hypertension,
  * Yes
  * NO Ischemic Heart Disease,
  * Yes
  * NO Dialysis
  * Yes
  * NO
Surgical procedure | Two days
  Specialty and type of intervention. Duration of the surgical intervention. Postoperative follow-up time hours
Vasoactive support | Two days
  Yes/Not, type quantity ml

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Bellvitge, L'Hospitalet de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
Approval of the study by the AEMPS and the CEIC of the Bellvitge University Hospital February - March 2018.
  Throughout this period of time, the promotion and inclusion of the different participating centers will be carried out. In addition to simultaneously performing the online database by the Statistics Department of the IDIBELL Foundation - Barcelona.
  Obtaining the approvals of the CEICS and relevant entities.
  It is expected that the days to make the cut can be done in February 2019.
  Subsequently, the statistical analysis will be carried out and the results will be presented at the Meeting of the Haemostasis, Transfusion Medicine and Fluid Therapy Section of the SEDAR in 2019 and the results will be sent to the journal that is deemed appropriate for publication.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: At the end of 2019
URL: http://fluidday.com

REFERENCES:
- [Background] Basora M, Colomina MJ, Moral V, Asuero de Lis MS, Boix E, Jover JL, Llau JV, Rodrigo MP, Ripolles J, Calvo Vecino JM. Clinical practice guide for the choice of perioperative volume-restoring fluid in adult patients undergoing non-cardiac surgery. Rev Esp Anestesiol Reanim. 2016 Jan;63(1):29-47. doi: 10.1016/j.redar.2015.06.013. Epub 2015 Sep 3. English, Spanish. PMID 26343809
- [Background] Colomina MJ, Basora M, Moral V, Llau JV. Crystalloids and hydroxyethyl starches in noncardiac surgical patients. Eur J Anaesthesiol. 2017 Jan;34(1):28-29. doi: 10.1097/EJA.0000000000000464. No abstract available. PMID 27136489
- [Background] Calvo-Vecino JM, Ripolles-Melchor J, Mythen MG, Casans-Frances R, Balik A, Artacho JP, Martinez-Hurtado E, Serrano Romero A, Fernandez Perez C, Asuero de Lis S; FEDORA Trial Investigators Group. Effect of goal-directed haemodynamic therapy on postoperative complications in low-moderate risk surgical patients: a multicentre randomised controlled trial (FEDORA trial). Br J Anaesth. 2018 Apr;120(4):734-744. doi: 10.1016/j.bja.2017.12.018. Epub 2018 Feb 3. PMID 29576114
- [Background] Ripolles-Melchor J, Aldecoa C. Goal-directed Hemodynamic Therapy: Neither for Anyone, Neither the Same for Everyone. Anesthesiology. 2018 Mar;128(3):682-683. doi: 10.1097/ALN.0000000000002050. No abstract available. PMID 29438252
- [Background] Ripolles-Melchor J, Chappell D, Aya HD, Espinosa A, Mythen MG, Abad-Gurumeta A, Bergese SD, Casans-Frances R, Calvo-Vecino JM. Erratum to: "Fluid therapy recommendations for major abdominal surgery. Via RICA recommendations revisited. Part III: Goal directed hemodynamic therapy. Rationale for maintaining vascular tone and contractility" [Rev Esp Anestesiol Reanim. 2017;64(6):348-359]. Rev Esp Anestesiol Reanim. 2017 Aug-Sep;64(7):425. doi: 10.1016/j.redar.2017.06.004. No abstract available. English, Spanish. PMID 28709478
- [Background] Ripolles-Melchor J, Chappell D, Aya HD, Espinosa A, Mythen MG, Abad-Gurumeta A, Bergese SD, Casans-Frances R, Calvo-Vecino JM. Erratum to: "Fluid therapy recommendations for major abdominal surgery. Via RICA recommendations revisited. Part II: Goal directed hemodynamic therapy. Rationale for optimising intravascular volume" [Rev Esp Anestesiol Reanim. 2017;64(6):339-347]. Rev Esp Anestesiol Reanim. 2017 Aug-Sep;64(7):424. doi: 10.1016/j.redar.2017.06.003. No abstract available. English, Spanish. PMID 28709477
- [Background] Ripolles-Melchor J, Chappell D, Espinosa A, Mythen MG, Abad-Gurumeta A, Bergese SD, Casans-Frances R, Calvo-Vecino JM. Erratum to: "Perioperative fluid therapy recommendations for major abdominal surgery. Via RICA recommendations revisited. Part I: Physiological background" [Rev Esp Anestesiol Reanim. 2017;64(6):328-338]. Rev Esp Anestesiol Reanim. 2017 Aug-Sep;64(7):423. doi: 10.1016/j.redar.2017.06.002. No abstract available. English, Spanish. PMID 28709476
- [Background] Ripolles-Melchor J, Chappell D, Espinosa A, Mhyten MG, Abad-Gurumeta A, Bergese SD, Casans-Frances R, Calvo-Vecino JM. Perioperative fluid therapy recommendations for major abdominal surgery. Via RICA recommendations revisited. Part I: Physiological background. Rev Esp Anestesiol Reanim. 2017 Jun-Jul;64(6):328-338. doi: 10.1016/j.redar.2017.02.008. Epub 2017 Mar 30. No abstract available. English, Spanish. PMID 28364973
- [Background] Ripolles-Melchor J, Chappell D, Aya HD, Espinosa A, Mhyten MG, Abad-Gurumeta A, Bergese SD, Casans-Frances R, Calvo-Vecino JM. Fluid therapy recommendations for major abdominal surgery. Via RICA recommendations revisited. Part II: Goal directed hemodynamic therapy. Rationale for optimising intravascular volume. Rev Esp Anestesiol Reanim. 2017 Jun-Jul;64(6):339-347. doi: 10.1016/j.redar.2017.02.009. Epub 2017 Mar 24. No abstract available. English, Spanish. PMID 28343684
- [Background] Ripolles-Melchor J, Chappell D, Aya HD, Espinosa A, Mhyten MG, Abad-Gurumeta A, Bergese SD, Casans-Frances R, Calvo-Vecino JM. Fluid therapy recommendations for major abdominal surgery. Via RICA recommendations revisited. Part III: Goal directed hemodynamic therapy. Rationale for maintaining vascular tone and contractility. Rev Esp Anestesiol Reanim. 2017 Jun-Jul;64(6):348-359. doi: 10.1016/j.redar.2017.03.002. Epub 2017 Mar 24. No abstract available. English, Spanish. PMID 28343682
- [Background] Ripolles-Melchor J, Alvarez-Baena L, Espinosa A, Calvo-Vecino JM. Preoperative fluid loading in major abdominal surgery. Eur J Anaesthesiol. 2017 Jan;34(1):43-44. doi: 10.1097/EJA.0000000000000512. No abstract available. PMID 27898485
- [Background] Ripolles Melchor J, Fries D, Chappell D. Colloidophobia. Minerva Anestesiol. 2016 Oct;82(10):1039-1042. Epub 2016 Jun 28. No abstract available. PMID 27352071
- [Background] Ripolles-Melchor J, Casans-Frances R, Espinosa A, Abad-Gurumeta A, Feldheiser A, Lopez-Timoneda F, Calvo-Vecino JM; EAR Group, Evidence Anesthesia Review Group. Goal directed hemodynamic therapy based in esophageal Doppler flow parameters: A systematic review, meta-analysis and trial sequential analysis. Rev Esp Anestesiol Reanim. 2016 Aug-Sep;63(7):384-405. doi: 10.1016/j.redar.2015.07.009. Epub 2016 Feb 10. English, Spanish. PMID 26873025
- [Background] Ripolles-Melchor J, Espinosa A, Martinez-Hurtado E, Abad-Gurumeta A, Casans-Frances R, Fernandez-Perez C, Lopez-Timoneda F, Calvo-Vecino JM. Perioperative goal-directed hemodynamic therapy in noncardiac surgery: a systematic review and meta-analysis. J Clin Anesth. 2016 Feb;28:105-15. doi: 10.1016/j.jclinane.2015.08.004. Epub 2015 Oct 2. PMID 26440438
- [Background] Cecconi M, Hofer C, Teboul JL, Pettila V, Wilkman E, Molnar Z, Della Rocca G, Aldecoa C, Artigas A, Jog S, Sander M, Spies C, Lefrant JY, De Backer D; FENICE Investigators; ESICM Trial Group. Fluid challenges in intensive care: the FENICE study: A global inception cohort study. Intensive Care Med. 2015 Sep;41(9):1529-37. doi: 10.1007/s00134-015-3850-x. Epub 2015 Jul 11. PMID 26162676
- [Background] Ripolles Melchor J, Espinosa A, Martinez Hurtado E, Casans Frances R, Navarro Perez R, Abad Gurumeta A, Calvo Vecino JM. Colloids versus crystalloids in the prevention of hypotension induced by spinal anesthesia in elective cesarean section. A systematic review and meta-analysis. Minerva Anestesiol. 2015 Sep;81(9):1019-30. Epub 2014 Dec 11. PMID 25501602
- [Background] Ripolles Melchor J, Espinosa A. [Goal directed fluid therapy controversies in non-cardiac surgery]. Rev Esp Anestesiol Reanim. 2014 Nov;61(9):477-80. doi: 10.1016/j.redar.2014.09.001. Epub 2014 Oct 3. No abstract available. Spanish. PMID 25284819
- [Background] Meier J, Filipescu D, Kozek-Langenecker S, Llau Pitarch J, Mallett S, Martus P, Matot I; ETPOS collaborators. Intraoperative transfusion practices in Europe. Br J Anaesth. 2016 Feb;116(2):255-61. doi: 10.1093/bja/aev456. PMID 26787795
- [Background] Caballo C, Escolar G, Diaz-Ricart M, Lopez-Vilchez I, Lozano M, Cid J, Pino M, Beltran J, Basora M, Pereira A, Galan AM. Impact of experimental haemodilution on platelet function, thrombin generation and clot firmness: effects of different coagulation factor concentrates. Blood Transfus. 2013 Jul;11(3):391-9. doi: 10.2450/2012.0034-12. Epub 2012 Sep 19. PMID 23058866
- [Background] Basora M, Moral V, Llau JV, Silva S. [Perioperative colloid administration: a survey of Spanish anesthesiologists' attitudes]. Rev Esp Anestesiol Reanim. 2007 Mar;54(3):162-8. Spanish. PMID 17436654
- [Background] Basora M, Llau JV. [Survey on the perioperative use of colloids]. Rev Esp Anestesiol Reanim. 2004 Oct;51(8):479. No abstract available. Spanish. PMID 15586550
- [Background] Llau JV, Acosta FJ, Escolar G, Fernandez-Mondejar E, Guasch E, Marco P, Paniagua P, Paramo JA, Quintana M, Torrabadella P. Multidisciplinary consensus document on the management of massive haemorrhage (HEMOMAS document). Med Intensiva. 2015 Nov;39(8):483-504. doi: 10.1016/j.medin.2015.05.002. Epub 2015 Jul 29. English, Spanish. PMID 26233588
- [Background] Guilabert P, Usua G, Martin N, Abarca L, Barret JP, Colomina MJ. Fluid resuscitation management in patients with burns: update. Br J Anaesth. 2016 Sep;117(3):284-96. doi: 10.1093/bja/aew266. PMID 27543523
- [Background] Guilabert P, Abarca L, Martin N, Usua G, Barret JP, Colomina MJ. What about HES in burn patients?: Evaluation of the actual evidence. Burns. 2018 May;44(3):489-493. doi: 10.1016/j.burns.2017.09.023. Epub 2017 Oct 10. No abstract available. PMID 29029856
- [Derived] Colomina MJ, Ripolles-Melchor J, Guilabert P, Jover JL, Basora M, Cassinello C, Ferrandis R, Llau JV, Penafiel J. Observational study on fluid therapy management in surgical adult patients. BMC Anesthesiol. 2021 Dec 13;21(1):316. doi: 10.1186/s12871-021-01518-z. PMID 34903176
- Available data/document: web page — http://fluidday.com